NUS-IRB Reference Code: NUS-IRB-2024-259 [PWCI]
Protocol title: Exploring and Evaluating the Impact of 'Refresh and Reconnect!': A Museum based Heritage Programme for Older Persons with Cognitive Impairment [ReCognition Study]

Date of Document: 20 Jan 2025

Version No: 1  Date of Revision: 19 Dec 2024



## PARTICIPANT INFORMATION SHEET

You are invited to participate in a research study. This information sheet provides you with information about the research study. Where "personal data" is used, it means data about you which makes you identifiable: (i) from such data or (ii) from such data and other information which the National University of Singapore (NUS) has or is likely to have. The Principal Investigator (the research doctor or the person in charge of this research) or his/her representative will also describe this research to you and answer all your questions. Read the information below and ask questions about anything you don't understand before deciding whether or not to take part.

## **PART I: General Information**

NUS-IRB Reference Code: NUS-IRB-2024-259 [PWCI]

#### 1. Protocol title:

Exploring and Evaluating the Impact of 'Refresh and Reconnect!': A Museum-based Heritage Programme for Older Persons with Cognitive Impairment [ReCognition Study]

#### 2. Principal Investigator:

Dr Ad Maulod

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 6516 8344

E-mail: ad.maulod@duke-nus.edu.sg

#### Co-Investigators:

A/Prof Rahul Malhotra

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 6516 6721

E-mail: rahul.malhotra@duke-nus.edu.sg

Ms Sasha Rouse

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 65161901

E-mail: sasha@duke-nus.edu.sg

Mr Malcolm Ravindran

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 6601 2578

E-mail: malcolmr@duke-nus.edu.sg

Mr Yunjie Wong

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 6601 8148

E-mail: <a href="mailto:yunjie@duke-nus.edu.sg">yunjie@duke-nus.edu.sg</a>

#### 3. Whom should I call if I have any questions or problems?

Please contact the Principal Investigator, Dr. Ad Maulod, at 65168344 or ad.maulod@duke-nus.edu.sg for all research-related matters, and in the event of research-related injuries.

 Version No: 1
Date of Revision: 19 Dec 2024

This study has undergone an ethics review by the National University of Singapore Institutional Review Board (NUS-IRB). For an independent opinion specifically regarding the rights and welfare of research participants, you may contact a staff member of the National University of Singapore Institutional Review Board at telephone (+65) 6516 1234 IMondays to Thursdays from 8.30am to 6pm, and Fridays from 8.30am to 5.30pm, except public holidays] or email at irb@nus.edu.sg.

### Who can participate in the research? What is the expected duration of my participation? What is the duration of this research?

By registering to participate in the 'Refresh and Reconnect!' (R&R!) programme by the National Museum of Singapore, you are invited to participate in a study to evaluate the efficacy of the R&R! programme. Eligible participants must meet the following criteria:

- Fulfil the 'Refresh and Reconnect!' recruitment criteria; and registers to participate in the programme;
- Willing and able to participate in surveys or interviews independently without proxy;
- Has score on the Montreal Cognitive Assessment (MoCA) screener ranging from 22 to 27 (if you have 10 or more years of education) OR 22 to 26 (if you have had less than 10 years of education)
- Do not have an existing diagnosis of moderate or severe dementia

Your involvement in this study is expected to last for no more than a period of 6 months. During this time, you are expected to participate in the 6-week R&R! programme at National Museum of Singapore, for a total of 6 visits (once weekly), each lasting approximately 2 hours, to the National Museum of Singapore.

#### 5. What is the approximate number of research subjects involved?

Up to 120 participants are expected to be involved in the programme, ethnographic observations and the quantitative component of this study. Up to 16 participants may be selected to be involved in the subsequent qualitative in-depth interviews for this study.

#### 6. What will be done if I take part in this research study?

R&R! Programme: If you consent to participate in this study, you are expected to take part in all sessions (where possible) of the 'Refresh and Reconnect!' programme hosted by the National Museum of Singapore. During this programme, you will participate in a 2hour weekly session over an 6-week period which includes guided tours of the National Museum and artist-led hands-on activities based on various art forms (for example, music and movement, handicraft, storytelling). At the end of each session, you will be asked to fill in a short 12-question survey which assesses your feelings about the programme, lasting approximately 5 minutes.

Ethnographic Observations: During the course of your participation in the R&R! programme, researchers may be present on-site to observe the conduct of the programme. Members of the study team may have open, informal conversations with you or your accompanying caregivers to gather your feedback about the programme, or to understand more about you. You may decline to be personally engaged by the study team in conversations, or you may decline answering their questions. You may, however, still be engaged if you are present in a group setting with other participants who have consented to be spoken to.

With your permission, specific photos or video clips may be taken by the research team during the visits, strictly to supplement the notes taken in documenting observations and insights. Photography and videography will be limited to capturing the museum space, and the R&R! programme; if persons are included in the frame of the photos/videos, the research team will ensure to take wide angle, side or back shots. We will not take any identifiable photos and videos, or those that contain sensitive information (e.g., personal photos within the centre) without your expressed consent. Where you did not give consent for photography or videography but happen to be captured in any photograph or video, the study team will mask your face or any identifiable features (E.g. blurring, mosaic).

> Version No: 1  Date of Revision: 19 Dec 2024

Quantitative Surveys: You are also expected to complete two surveys, each survey is expected to last between no more than 1 hour. The pre-programme baseline assessment will be conducted approximately up to 4 weeks prior to your participation in the R&R! programme, and the post-programme assessment will be conducted approximately 1 to 2 weeks after completion of the programme.

The survey questionnaire includes measurement of your cognitive status, general and health-related quality of life, presence or intensity of anxiety and depressive symptoms, loneliness level, and your motivations to learn.

You may take breaks during any of the surveys by notifying the member of the study team. You do not need to answer any questions that you do not wish to. Participation in this research study is voluntary.

Qualitative In-depth Interviews: If selected for this component of the study, you may be asked to take part in one semi-structured interview, lasting approximately 1 to 1.5 hours each. The *in-depth interview* takes place up to 1 month after completing the programme. You will be asked about your perception of the museum and towards heritage-based arts programmes, your perception of the 'Refresh and Reconnect!' programme, about your responses to the quantitative survey, and how the programme can be better for you.

You may take breaks during any interview session by notifying the interviewer. You do not need to answer any questions that you do not wish to. All sessions may be audiorecorded, with your consent. All audio-recorded sessions and written notes will be transcribed or typed out. We will not include any personal details in the transcript. If you agree, the notes from these sessions may also be used for future research.

Participation in this research study is voluntary, a member of the study team will contact you if you are invited to participate in the in-depth interviews. Non-participation in the indepth interviews will not affect your ability to participate in the R&R! programme or the surveys in any way.

#### 7. Will there be reimbursement for reasonable transport costs and time spent from my participation?

There will be a reimbursement of SGD40 upon completion of both quantitative surveys by you.

If you are recruited and complete the semi-structured interview, you will be reimbursed with an additional SGD30 in cash. Non-participation in this component of the research will not affect your reimbursement from completion of the quantitative surveys.

#### 8. How will my privacy and the confidentiality of my research records be protected?

NUS has established data management policies and rules for protection of the personal data of human research subjects in NUS studies, including the collection, use and storage of such data.

Additionally, our researchers are required to comply with the Human Biomedical Research Act (HBRA) and other applicable laws. Under the HBRA and the Personal Data Protection Act (PDPA), researchers must take all reasonable steps and safeguards as needed to protect individually identifiable information or material against accidental or unlawful loss, modification or destruction, or unauthorised access, disclosure, copying, use or modification.

For purposes of validating the research findings and supporting future research work, research data (without personal identifiers) used in any publication will be kept for a minimum of 10 years before being discarded in accordance with the NUS Research Data Management Policy.

>  Version No: 1 Date of Revision: 19 Dec 2024

## PART II: Information on this Human Biomedical Research

#### 9. What is the nature of this biomedical research?

This research is an exploratory study to evaluate the impact of a non-pharmaceutical, intervention on the health and well-being of persons with cognitive impairment. The interventions used in this research are under evaluation and are not currently validated as standard care or standard practice.

### What is the purpose of this biomedical research?

This study aims to explore and evaluate the impact of "Refresh and Reconnect!" (R&R!), a museum-based heritage programme launched by the National Museum of Singapore, on the health and well-being of persons with cognitive impairment.

Your participation may contribute to the understanding of how participation in the R&R! programme impacts the health and well-being of persons living with cognitive impairment (PWCIs), and their perception of the museum. Additionally, your participation may also provide insight into the factors, contexts, and mechanisms that influence the effect and implementation of the museum-based intervention, as well as to elucidate any placebased effects of the National Museum of Singapore's Reunion space.

## What are the possible risks, discomforts or inconveniences to me if I participate in this research?

You may experience some fatigue while responding to the questions in the surveys or interviews. If you find that some questions are distressful for you or are difficult to answer. please know that you do not have to answer any question that you do not wish to, and you can stop or postpone the interview at any point. You can also choose to terminate the interview indefinitely and/or withdraw from this research without repercussions. If you experience discomfort during the programme at any point, you may also choose to take a break by informing any member of the research team, or any staff member or volunteer from the National Museum of Singapore.

With your consent, specific photos or video clips may be taken by the research team during the ethnographic observations, strictly to supplement the notes taken in documenting observations and insights. Photography and videography will be limited to inanimate objects or spaces, and if persons are included, the research team will ensure to take wide angle, side or back shots. We will not take any identifiable photos and videos, or those that contain sensitive information (e.g., personal photos within the centre) without your expressed consent. Where you did not give consent for photography or videography but happen to be captured in any photograph or video, the study team will mask your face or any identifiable features (E.g. blurring, mosaic).

If you are selected for, and consent to participation in the in-depth interviews, the research team will seek your consent to audio-record interviews. If you do not consent to audiorecording for the in-depth interviews, members of the study team will instead take detailed notes of your responses.

#### 12. What benefits can I expect from participating in the research?

There is no direct benefit to you by participating in this research study. The knowledge gained may benefit the public in the future about the impact of museum-based programme such as 'Refresh and Reconnect!' for person living with cognitive impairment, from which the programme may improve for its future participants.

The program may offer you opportunities for social interactions between participants, museum staff, and volunteers, which may foster a sense of community and belonging during the programme.

>  Version No: 1 Date of Revision: 19 Dec 2024

# 13. Are there any alternative procedures or treatments available to me? What are the potential benefits and risks of such alternatives?

There are no alternative treatments for participants as this is not a scheduled procedure for cognitive impairment management.

# 14. If I am injured as a result of participating in this research, what are the compensation and treatments available to me?

If you follow the directions of the PI in charge of this research study and you are injured, NUS will pay the medical expenses for the treatment of that injury. By signing this consent form, you will not waive any of your legal rights or release the parties involved in this study from liability for negligence.

### 15. Do I have to incur any expenses by participating in this research?

There are no anticipated expenses that you will be expected to incur by participating in this research; transport to the National Museum of Singapore will be provided from the relevant site from which you are recruited from, if possible.

## 16. Will my participation in this research involve the use of any information that will identify me?

Participants' personal data (i.e. name and phone number) will be collected in this study for the purpose of contact for follow-up interviews and surveys only.

#### 17. How will my personal identifiers collected from me be kept confidential?

Only the principal investigator, co-investigators, and authorised study team members will have access to your personal data (e.g., names and contact number) on a need-to-know basis. This data will not be released to any other person, unless required by applicable laws and regulations e.g., Infectious Diseases Act. Your personal data will never be used in a publication or presentation. To protect your confidentiality, your data will to the extent feasible during the study, be anonymized or coded (i.e., only identified with a code number). All personal data (e.g., names and contact information) will be kept separate from the research data. The link between your personal data and the code number will be kept confidential by the principal investigator. In either case, we cannot reduce the risk to zero.

We will store all recorded audio/video of your interviews, transcripts and all survey responses on this study's Dropbox folder, a secure online server co-managed by NUS. Dropbox access to this study will only be given to the research team, and access is authenticated via two-factor authentication (2FA).

We will do our best to protect your data during storage and when they are shared. However, there remains a possibility that someone could identify you.

# 18. Will any identifiable information obtained from me be used for future biomedical research?

If you consent, your personal data (e.g., name and phone number) will be retained after the study so that we may re-contact you for participation in future research and/or follow-up procedures in this study.

## 19. Will I be re-identified in the event of incidental finding(s) arising during the biomedical research?

As there are no anticipated incidental findings that may be discovered in the course of this study, you will not be re-identified or notified.

### 20. Under what circumstances will I be re-contacted for further consent?

Should there be any changes in terms of your involvement in the study beyond the scope of research explained to you in this information sheet (e.g., study duration, cancellation

 Version No: 1
Date of Revision: 19 Dec 2024

of study), we will seek your further re-consent for your continued participation in this study.

### 21. Can I withdraw my consent to the research at any time?

You can withdraw from the research at any time without giving any reasons, by informing the principal investigator verbally or in writing. Please note that the withdrawal of consent does not affect the research information obtained before the consent is withdrawn and such information may still be retained and used for research. There will be no penalties or damages imposed on you should you withdraw your consent to participate in this research.

### 22. Will my personal data be shared and / or processed for use in research?

Your personal data may, for the purposes of use in this study, relevant laws and/ or the Singapore Government ("Research Studies"), be processed into anonymized or coded/de-identified data ("Anonymized/ De-identified Dataset"). Such processing may be done by us or with the assistance of our authorized data service providers or data intermediaries."

 Version No: 1
Date of Revision: 19 Dec 2024

## **Consent Form for Research Subjects**

#### Protocol title:

Exploring and Evaluating the Impact of 'Refresh and Reconnect!': A Museum-based Heritage Programme for Older Persons with Cognitive Impairment [ReCognition Study]

#### **Principal Investigator:**

Dr Ad Maulod

Centre for Ageing Research and Education, Duke-NUS Medical School 8 College Road Singapore 169857

Tel: 6516 8344

E-mail: ad.maulod@duke-nus.edu.sg

I hereby acknowledge that:

- My signature is my acknowledgement that I have agreed to take part in the above research.
- I have received a copy of this information sheet that explains the use of my data this research. I understand its contents and agree to donate my data for the use of this research. I confirm that I consent to the collection, use, disclosure and processing of my data for the purposes of the study.
- If I choose to withdraw from the study before it is completed, I agree to the continued use of my research data up to the time of my withdrawal, for this research. I understand that due to the nature of the ethnographic observations, it is impracticable to withdraw or destroy all research data collected for this component of the study. I am aware that that the withdrawal of consent does not affect the research information obtained before the consent is withdrawn and such information may still be retained and used for research.
- I consent / do not consent\* to have the coded data made available for future research studies. This will be subject to an Institutional Review Board's approval.
- I agree / do not agree\* to be re-contacted for future related studies. I understand that future studies will be subject to an Institutional Review Board's approval.
- I agree/ do not agree\* to the audio-recording/ photo-taking/ video-recording\* of my participation in the research. I understand that although my name will be not associated with the quotes/photographs/videorecordings used in publication/presentation, I may still be identified.

| ** This research has been explained to me in [state language), which I unders [name of translator] on [date). | tand, by |
|---|---|
| Name and Signature (Research Subject) | <br>Date |
| I, the undersigned, certify to the following: (a) I am 21 years of age or older. (b) I have taken reasonable steps to ascertain the identity of the research subject. (c) To the best of my knowledge, the research subject had the study fully explained in a language underst understands the nature, risks and benefits of his/ her participation in the study. (d) I have taken steps to ascertain that the consent has been given voluntarily without any coercion or in | |
| Name and Signature (Witness) | <br>Date |
| Name and Signature (Consent Taker) | <br>Date |
| **The study has been explained to the research subject in [State language] | |
| **Name and Signature (Translator) | <br>Date |

## NUS-IRB Reference Code: NUS-IRB-2024-259 [Artist/Staff]

**Protocol title:** Exploring and Evaluating the Impact of 'Refresh and Reconnect!': A Museum based Heritage Programme for Older Persons with Cognitive Impairment [ReCognition Study]

Date of Document: 20 Jan 2025

 Version No: 1
Date of Revision: 19 Dec 2024



### PARTICIPANT INFORMATION SHEET

You are invited to participate in a research study. This information sheet provides you with information about the research study. Where "personal data" is used, it means data about you which makes you identifiable: (i) from such data or (ii) from such data and other information which the National University of Singapore (NUS) has or is likely to have. The Principal Investigator (the research doctor or the person in charge of this research) or his/her representative will also describe this research to you and answer all your questions. Read the information below and ask questions about anything you don't understand before deciding whether or not to take part.

## **PART I: General Information**

NUS-IRB Reference Code: NUS-IRB-2024-259 [Artist/Staff]

#### 1. Protocol title:

Exploring and Evaluating the Impact of 'Refresh and Reconnect!': A Museum-based Heritage Programme for Older Persons with Cognitive Impairment [ReCognition Study]

#### 2. Principal Investigator:

Dr Ad Maulod

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 6516 8344

E-mail: ad.maulod@duke-nus.edu.sg

### **Co-Investigators:**

A/Prof Rahul Malhotra

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 6516 6721

E-mail: rahul.malhotra@duke-nus.edu.sg

Ms Sasha Rouse

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 65161901

E-mail: sasha@duke-nus.edu.sg

Mr Malcolm Ravindran

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 6601 2578

E-mail: malcolmr@duke-nus.edu.sg

Mr Yunjie Wong

Centre for Ageing Research and Education, Duke-NUS Medical School

8 College Road Singapore 169857

Tel: 6601 8148

E-mail: yunjie@duke-nus.edu.sg

#### 3. Whom should I call if I have any questions or problems?

Please contact the Principal Investigator, Dr. Ad Maulod, at 65168344 or ad.maulod@duke-nus.edu.sg for all research-related matters, and in the event of research-related injuries.

 Version No: 1
Date of Revision: 19 Dec 2024

This study has undergone an ethics review by the National University of Singapore Institutional Review Board (NUS-IRB). For an independent opinion specifically regarding the rights and welfare of research participants, you may contact a staff member of the National University of Singapore Institutional Review Board at telephone (+65) 6516 1234 [Mondays to Thursdays from 8.30am to 6pm, and Fridays from 8.30am to 5.30pm, except public holidays] or email at irb@nus.edu.sg.

#### 4. Who can participate in the research? What is the expected duration of my participation? What is the duration of this research?

You have been invited to take part in the qualitative component of the ReCognition study because you are either a museum staff who has been involved in coordinating or planning the 'Refresh & Reconnect!' (R&R) programme, or you are an artist who has hosted one or more of the sections of the R&R programme. Eligible participants must meet the following criteria:

- Is a museum staff who works part-time or full-time with National Museum of Singapore, and coordinated in at least one out of eight runs of R&R program OR
- Is an artist who worked with the National Museum of Singapore to lead or facilitate one of the sections for the R&R! program
- Is able to respond to interviews independently

Your involvement in this study will take place alongside your involvement in the R&R! programme. Museum staff will be interviewed during their time working with the programme. All artists involving in the programme will be interviewed during their time working with the programme. Interviews may be conducted as part of the ethnographic observations component of the study, or a member of the study team may request to speak to you in a separate session, with your consent.

Ethnographic observations will take place during the 2-hour R&R! programme. Ethnographic interviews, where necessary, are expected to last no longer than 1.5 hours.

#### 5. What is the approximate number of research subjects involved? Three museum staff and six participating artists are expected to be involved in the programme, ethnographic observations and the qualitative component of this study.

#### 6. What will be done if I take part in this research study?

#### Museum staff of R&R!

Ethnographic Observations: During the course of your participation in the R&R! programme, researchers may be present on-site to observe the conduct of the programme. Members of the study team may ask you questions or informally converse with you in order to find out more about your role in facilitating the R&R! programme, as well as to understand the objectives and challenges in facilitating the programme further.

Ethnographic unstructured Interviews: In this component of the study, you may be asked to take part in two unstructured interviews. The pre-programme interview will take place approximately before the start, or at the start of your involvement in the R&R! programme for this study period; the post-programme interviews take place towards the conclusion of the study period, or at the end of your involvement in the R&R! programme. At the pre-programme interview, you will be asked about your processes, motivations and objectives of designing museum-based interventions for PWCIs, including outreach efforts, programme expectations and perceptions of 'success'. At the post-programme interview, you will be asked for feedback about each session, and programme enablers and barriers that may impact the programme.

#### **Artist of R&R!**

Ethnographic Observations: During the course of your facilitating or conducting the R&R! programme, researchers may be present on-site to observe the conduct of the programme. Members of the study team may ask you questions or informally converse with you in order to find out more about your involvement in the R&R! programme as well as to understand the objectives and challenges in facilitating the programme further

Qualitative In-depth Interviews: You will be asked to take part in several short unstructured interviews, conducted throughout the overall programme segment for which you are involved. You will be asked about your programme vision and previous exposure with curating programmes for older persons and experiences working with both the programme organisers, PWCIs as well as volunteers and accompanying caregivers, your experience conducting the programme, and enablers and barriers that may impact the programme. Members of the study team may request to speak to you on a separate occasion, outside of the R&R! programme segment, with your consent.

#### For all participants

With your permission, specific photos or video clips may be taken by the research team during the visits, strictly to supplement the notes taken in documenting observations and insights. Photography and videography will be limited to capturing the museum space, and the R&R! programme; if persons are included in the frame of the photos/videos, the research team will ensure to take wide angle, side or back shots. We will not take any identifiable photos and videos, or those that contain sensitive information (e.g., personal photos within the centre) without your expressed consent. Where you did not give consent for photography or videography but happen to be captured in any photograph or video, the study team will mask your face or any identifiable features (E.g. blurring, mosaic).

You may take breaks during any interview session by notifying the interviewer. You do not need to answer any questions that you do not wish to. Interviews may be audiorecorded, with your consent. All audio-recorded sessions and written notes will be transcribed or typed out. We will not include any personal details in the transcript. If you agree, the notes from these sessions may also be used for future research. Participation in this research study is voluntary; however, due to the ethnographic observations, members of the research team will be present on-site to observe the conduct of the R&R! programme regardless of your participation in this component of the study.

#### 7. Will there be reimbursement for reasonable transport costs and time spent from my participation?

There will be a reimbursement of SGD50 in cash upon completion of unstructured interviews for artists. There is no reimbursement for museum staff who complete this component of the study.

#### 8. How will my privacy and the confidentiality of my research records be protected?

NUS has established data management policies and rules for protection of the personal data of human research subjects in NUS studies, including the collection, use and storage of such data.

Additionally, our researchers are required to comply with the Human Biomedical Research Act (HBRA) and other applicable laws. Under the HBRA and the Personal Data Protection Act (PDPA), researchers must take all reasonable steps and safeguards as needed to protect individually identifiable information or material against accidental or unlawful loss, modification or destruction, or unauthorised access, disclosure, copying, use or modification.

For purposes of validating the research findings and supporting future research work, research data (without personal identifiers) used in any publication will be kept for a minimum of 10 years before being discarded in accordance with the NUS Research Data Management Policy.

## PART II: Information on this Human Biomedical Research

#### 9. What is the nature of this biomedical research?

This research is an exploratory study to evaluate the impact of a non-pharmaceutical, intervention on the health and well-being of persons with cognitive impairment. The interventions used in this research are under evaluation and are not currently validated as standard care or standard practice.

### 10. What is the purpose of this biomedical research?

This study aims to explore and evaluate the impact of "Refresh and Reconnect!" (R&R!), a museum-based heritage programme launched by the National Museum of Singapore, on the health and well-being of persons with cognitive impairment.

Your participation may also provide insight into the factors, contexts, and mechanisms that influence the effect and implementation of the museum-based intervention. Additionally, your participation could benefit the quality of future runs of the R&R! programme.

# 11. What are the possible risks, discomforts or inconveniences to me if I participate in this research?

You may experience some fatigue while responding to the questions in the interviews. If you find that some questions are distressful for you or are difficult to answer, please know that you do not have to answer **any** question that you do not wish to, and you can stop or postpone the interview at any point. You may also choose to take breaks at any point during the interview. You can also choose to terminate the interview indefinitely and/or withdraw from this research without repercussions.

With your consent, specific photos or video clips may be taken by the research team during the ethnographic observations, strictly to supplement the notes taken in documenting observations and insights. Photography and videography will be limited to inanimate objects or spaces, and if persons are included, the research team will ensure to take wide angle, side or back shots. We will not take any identifiable photos and videos, or those that contain sensitive information (e.g., personal photos within the centre) without your expressed consent. Where you did not give consent for photography or videography but happen to be captured in any photograph or video, the study team will mask your face or any identifiable features (E.g. blurring, mosaic). The research team will also seek your consent to audio-record interviews. If you do not consent to audio-recording for the in-depth interviews, members of the study team will instead take detailed notes of your responses.

#### 12. What benefits can I expect from participating in the research?

There is no direct benefit to you as an individual by participating in this research study. Knowledge that you gain from participating in the research could help you better understand the facilitators of R&R! programme success.

The knowledge gained may benefit the public in the future about the impact of museum-based program such as 'Refresh and Reconnect!' for person living with cognitive impairment, from which the programme may improve for its future participants.

# 13. Are there any alternative procedures or treatments available to me? What are the potential benefits and risks of such alternatives?

There are no alternative treatments for participants. Participation in this study is, however, voluntary and not providing consent will have no impact on your involvement in the R&R! programme nor on any other aspect of your work.

 Version No: 1
Date of Revision: 19 Dec 2024

# 14. If I am injured as a result of participating in this research, what are the compensation and treatments available to me?

If you follow the directions of the PI in charge of this research study and you are injured, NUS will pay the medical expenses for the treatment of that injury. By signing this consent form, you will not waive any of your legal rights or release the parties involved in this study from liability for negligence.

### 15. Do I have to incur any expenses by participating in this research?

There are no anticipated expenses that you will incur as a consequence of your participation in this research study.

# 16. Will my participation in this research involve the use of any information that will identify me?

Participants' personal data (i.e. name and phone number) will be collected in this study for the purpose of contact for follow-up interviews only.

## 17. How will my personal identifiers collected from me be kept confidential?

Only the principal investigator, co-investigators, and authorised study team members will have access to your personal data (e.g., names and contact number) on a need-to-know basis. This data will not be released to any other person, unless required by applicable laws and regulations e.g., Infectious Diseases Act. Your personal data will never be used in a publication or presentation. To protect your confidentiality, your data will to the extent feasible during the study, be anonymized or coded (i.e., only identified with a code number). All personal data (e.g., names and contact information) will be kept separate from the research data. The link between your personal data and the code number will be kept confidential by the principal investigator. In either case, we cannot reduce the risk to zero.

We will store all recorded audio/video of your interviews, and transcripts on this study's Dropbox folder, a secure online server co-managed by NUS. Dropbox access to this study will only be given to the research team, and access is authenticated via two-factor authentication (2FA). Audio-recordings from the interview will be destroyed after being transcribed and verified for accuracy by the study team.

We will do our best to protect your data during storage and when they are shared. However, there remains a possibility that someone could identify you.

# 18. Will any identifiable information obtained from me be used for future biomedical research?

If you consent, your personal data (e.g., name and phone number) will be retained after the study so that we may re-contact you for participation in future research and/or follow-up procedures in this study.

# 19. Will I be re-identified in the event of incidental finding(s) arising during the biomedical research?

As there are no anticipated incidental findings that may be discovered in the course of this study, you will not be re-identified or notified.

#### 20. Under what circumstances will I be re-contacted for further consent?

Should there be any changes in terms of your involvement in the study beyond the scope of research explained to you in this information sheet (e.g., study duration, cancellation of study), we will seek your further re-consent for your continued participation in this study.

#### 21. Can I withdraw my consent to the research at any time?

You can withdraw from the research at any time without giving any reasons, by informing the principal investigator verbally or in writing. Please note that the withdrawal of consent does not affect the research information obtained before the consent is withdrawn and such information may still be retained and used for research. There will be no penalties or damages imposed on you should you withdraw your consent to participate in this research.

#### 22. Will my personal data be shared and / or processed for use in research?

Your personal data may, for the purposes of use in this study, relevant laws and/ or the Singapore Government ("Research Studies"), be processed into anonymized or coded/de-identified data ("Anonymized/ De-identified Dataset"). Such processing may be done by us or with the assistance of our authorized data service providers or data intermediaries.

## **Consent Form for Research Subjects**

#### Protocol title:

Exploring and Evaluating the Impact of 'Refresh and Reconnect!': A Museum-based Heritage Programme for Older Persons with Cognitive Impairment [ReCognition Study] [Artist/Staff]

### **Principal Investigator:**

Dr Ad Maulod

Centre for Ageing Research and Education, Duke-NUS Medical School 8 College Road Singapore 169857

Tel: 6516 8344

Tel: 65 16 8344

e-mail: ad.maulod@duke-nus.edu.sg

I hereby acknowledge that:

- 1. My signature is my acknowledgement that I have agreed to take part in the above research.
- 2. I have received a copy of this information sheet that explains the use of my data this research. I understand its contents and agree to donate my data for the use of this research. I confirm that I consent to the collection, use, disclosure and processing of my data for the purposes of the study.
- 3. If I choose to withdraw from the study before it is completed, I agree to the continued use of my research data up to the time of my withdrawal, for this research. I understand that due to the nature of the ethnographic observations, it is impracticable to withdraw or destroy all research data collected for this component of the study. I am aware that that the withdrawal of consent does not affect the research information obtained before the consent is withdrawn and such information may still be retained and used for research."
- 4. I consent / do not consent\* to have the coded data made available for future research studies. This will be subject to an Institutional Review Board's approval.
- 5. I agree / do not agree\* to be re-contacted for future related studies. I understand that future studies will be subject to an Institutional Review Board's approval.
- 6. I agree/ do not agree\* to the audio-recording/ photo-taking/ video-recording\* of my participation in the research. I understand that although my name will be not associated with the quotes/photographs/video-recordings used in publication/presentation, I may still be identified.

| ** This | | hich I understand, by |
|---|---|---|
| | (name of translator) on (date). | |
| <br>Name | and Signature (Research Subject) | <br>Date |
| l tha | adorsioned portify to the following: | |
| i, trie u<br>(a) | ndersigned, certify to the following: I am 21 years of age or older. | |
| (b) | I have taken reasonable steps to ascertain the identity of the research subject. | |
| (c) | To the best of my knowledge, the research subject had the study fully explained in a | anguage understood by |
| ` , | him/ her and clearly understands the nature, risks and benefits of his/ her participation i | n the study. |
| (d) | I have taken steps to ascertain that the consent has been given voluntarily without any | coercion or intimidation. |
| <br>Name | and Signature (Witness) | Date |
| ———<br>Name | and Signature (Consent Taker) | <br>Date |
| | , | |
| **The s | study has been explained to the research subject in [State language] | |
| **Nam | ne and Signature (Translator) | Date |

 Version No: 1
Date of Revision: 19 Dec 2024